CLINICAL TRIAL: NCT06514534
Title: A Phase II, Multi-center, Prospective, Open-label Study of Asciminib in Patients With Chronic Myeloid Leukemia in Chronic Phase (CML-CP) or Accelerated Phase (CML-AP) With T315I Mutation Who Are Resistant, Intolerant or Ineligible to Ponatinib.
Brief Title: Open-label Study of Asciminib for CML-CP or CML-AP Patients With T315I Mutation Who Are Resistant, Intolerant or Ineligible to Ponatinib.
Acronym: ASC4TARGET
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CABL001AFR05; 2024-516049-38-00 (Registry Identifier: CTIS (EU) Number)
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Chronic Myeloid Leukemia (CML)
Keywords: Asciminib; ABL001; Abelson proto-oncogene (ABL1); Chronic Myelogenous Leukemia (CML); BCR::ABL1; Phase II; Tyrosine kinase inhibitor (TKI)
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — asciminib

STUDY DESIGN:
Intervention Model Description: Single-arm, open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Asciminib (Scemblix®) (Experimental): Asciminib will be administered 200 mg twice a day orally. The minimum dose is 200 mg, and maximum dose is 400 mg.
  Interventions: Drug: ABL001/Asciminib

INTERVENTIONS:
Drug: ABL001/Asciminib — The study treatment for this clinical trial is an investigational drug called asciminib, which is marketed under the brand name Scemblix®. Asciminib is a compound that is being evaluated for its efficacy and safety in the treatment of the target condition.
  The minimum dose of asciminib to be administered in this study is 200 mg, while the maximum dose is 400 mg. The dose is planned as 200 mg twice a day (BID).
  The drug will be administered orally, allowing for convenient and non-invasive administration.

SUMMARY:
The objective of this Phase II study is to assess the potential of asciminib in managing CML-CP or CML-AP in patient carrying the T315I mutation. The presence of this mutation introduces treatment difficulties due to the limited available options. The study seeks to collect additional data on the effectiveness and safety of asciminib for these patients. By determining the drug's capacity to manage the disease and enhance patients outcomes, the study is designed to fill the unmet medical need and potentially offer a new therapeutic path for patients at a treatment deadlock.

DETAILED DESCRIPTION:
This study is a Phase II, multi-center, single-arm prospective, open-label study that aims to evaluate the efficacy and safety of oral asciminib in patients with CML-CP or CML-AP with T315I mutation and after at least one tyrosine kinase inhibitors (TKI) and are resistant, intolerant, or ineligible for treatment with ponatinib.

Patients who have not been previously treated with asciminib would be enrolled in this study. The researchers will assess the effectiveness of asciminib in these participants, as well as evaluate its safety profile. The study will consist of two phases:

* The "core phase" which aims to answer the scientific and medical objectives.
* An "extension phase" intended to provide opportunity to the participants to continue their ongoing treatment (asciminib) up to commercialization in France or decision to not commercialize asciminib for the study population (stopping development, refusal to extend marketing authorization, refusal of reimbursement).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study.
* Male or female participants with a diagnosis of CML-CP or CML-AP ≥ 18 years of age.
* Patients with CML-CP or CML-AP with history of documented T315I mutation after at least one TKI and are resistant, intolerant, or ineligible to ponatinib (according to Investigator judgment)
* Not already treated with asciminib or another any allosteric TKI
* Failure (adapted from the 2020 & 2013 ELN Guidelines) or intolerance to Ponatinib at the time of Screening.
* Ineligible to ponatinib according to Investigator (based on EU ponatinib SmPC)
* Evidence of typical BCR::ABL1 transcript or atypical transcripts at the time of Screening which are amenable to standardized or non-standardized RQ-PCR quantification.

Exclusion Criteria:

* Previous hematopoietic allogeneic stem-cell transplantation
* Cardiac or cardiac repolarization abnormality
* Severe and/or uncontrolled concurrent medical disease that in the opinion of the Investigator could cause unacceptable safety risks or compromise compliance with the protocol (e.g. uncontrolled diabetes, active or uncontrolled infection, pulmonary hypertension)
* History of clinical acute pancreatitis within 1 year of study entry or past medical history of chronic pancreatitis (except if ponatinib-induced and completely resolved at time of Screening)
* History of acute or chronic liver disease (i.e., cirrhosis; liver impairment)
* Known presence of significant congenital or acquired bleeding disorder unrelated to cancer
* History of other active malignancy within 3 years prior to study entry with the exception of previous or concomitant basal cell skin cancer and previous carcinoma in situ treated curatively
* Known history of Human Immunodeficiency Virus (HIV), chronic Hepatitis B Virus (HBV), or chronic Hepatitis C Virus (HCV) infection. Testing for Hepatitis B surface antigen (HBs Ag) and Hepatitis B core antibody (HBcAb / anti HBc) will be performed at Screening
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection, or gastric bypass surgery)
* Treatment with medications that meet one of the following criteria and that cannot be discontinued at least one week prior to the start of treatment with study treatment:

  * Moderate or strong inducers of CYP3A
  * Moderate or strong inhibitors of CYP3A
* Pregnant or nursing (lactating) women
* Women of child-bearing potential
* Compound mutant T315I resistant to asciminib monotherapy (polyclonal ABL1 mutations including T315I can be enrolled) Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Rate of BCR::ABL1 (Breakpoint Cluster Region Gene::Abelson proto-oncogene) IS (International Scale) ≤ 1% [MR2 (Molecular Response 2)] | Month 12
  Evaluation of asciminib efficacy : proportion of patients with MR2 (BCR::ABL1 IS ≤1%) level of response at 12 months.

SECONDARY OUTCOMES:
Kinetics of response: BCR::ABL1 IS (MR2, MMR, MR4.0, MR4.5, undetectable MR4.5) | At 3, 6, 9, 12, 18 and 24 months
  Proportion of patients achieving the response levels (MR2, MMR, MR4.0, MR4.5, undetectable MR4.5)
Estimate response to treatment MR2 at 12 months in participants with BCR::ABL1 IS > 1% at treatment initiation or maintenance of MR2 at 12 months in participants with MR2 at treatment initiation | At 12 months
  Proportion of patients with MR2 level of response (BCR::ABL1 IS ≤ 1%) in participants without MR2 at treatment initiation or maintenance of MR2 at 12 months in participants with MR2 at treatment initiation.
Time to Major Molecular Response (MMR) (for participants not in MMR at treatment initiation) | up to 24 months
  Major Molecular Response (MMR) criteria is defined as a ≥ 3.0 log reduction in BCR::ABL1 transcripts compared to the standardized Baseline equivalent to ≤ 0.1 % BCR::ABL1 % by international scale as measured by RQ-PCR, confirmed by duplicate analysis of the same sample.
Duration of MMR | up to 24 months
  MMR criteria is defined as a ≥ 3.0 log reduction in BCR::ABL1 transcripts compared to the standardized Baseline equivalent to ≤ 0.1 % BCR::ABL1 % by international scale as measured by RQ-PCR, confirmed by duplicate analysis of the same sample.
Time to Molecular Response 2 (MR2) (for participants not in MR2 at treatment initiation) | up to 24 months
  MR2 criteria is defined as a ≥ 2.0 log reduction in BCR::ABL1 transcripts compared to the standardized Baseline equivalent to ≤ 1 % BCR::ABL1 % by international scale as measured by RQ-PCR, confirmed by duplicate analysis of the same sample.
Duration of MR2 | up to 24 months
  MR2 criteria is defined as a ≥ 2.0 log reduction in BCR::ABL1 transcripts compared to the standardized Baseline equivalent to ≤ 1 % BCR::ABL1 % by international scale as measured by RQ-PCR, confirmed by duplicate analysis of the same sample
Overall survival (OS) | up to 24 months
  Overall Survival (OS) is defined as the time from the first dose of study medication to death due to any cause. If a patient is not known to have died, then OS will be censored at the latest date the patient was known to be alive (on or before the cut-off date).
Progression Free Survival (PFS) | up to 24 months
  Progression Free Survival (PFS) is defined as time from the first dose of study medication to earliest occurrence of documented disease progression to AP/BC (depending on CML phase at asciminib initiation: CP or AP) or death due to any cause, whichever occurs first.
Event Free Survival (EFS) | up to 24 months
  Event Free Survival is defined as time from the first dose of study medication to an event which may include:
  * Treatment failure
  * Confirmed loss of MR2 at any time while on study treatment,
  * Discontinuation of study treatment due to AE,
  * Progression to AP/BC (including progressions observed during the survival follow up period),
  * Death from any cause (including deaths observed during the survival follow-up period).
Failure Free Survival (FFS) | up to 24 months
  Failure Free Survival (FFS) is defined as time from the first dose of study medication to a failure event which may include:
  * Treatment failure
  * Confirmed loss of MR2 at any time while on study treatment,
  * Discontinuation of study treatment due to AE.
Adverse events (AEs) and Serious Adverse events (SAEs) | up to 24 months
  Description/severity (grade of severity) of AE (all AE, serious or not serious AE, related and not related AE), and number of patients who discontinued the treatment due to AE.
Deaths and reasons for death | up to 24 months
  To evaluate the safety and tolerability profile of asciminib.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- France (2):
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Nantes

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.